CLINICAL TRIAL: NCT05239949
Title: Effects of Hypopressive Exercises in Comparison With Routine Pelvic Floor Exercises in Women With Urinary Incontinence: A Randomized Controlled Trial
Brief Title: Effects of Hypopressive Exercises in Comparison With Routine Pelvic Floor Exercises in Women With Urinary Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC-FSD-00282
Record Dates: First submitted 2022-02-04; First posted 2022-02-15 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Urinary Incontinence
Keywords: Urinary Incontinence; Pelvic floor exercises; Hypopressive exercises
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: our study will be single-blinded, outcome assessor will be blinded to avoid being biased during outcome assessment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypopressive exercises and electrical muscle stimulation (EMS) (Experimental): Women included in this group underwent 24 sessions during 8 weeks (3 days/ week). Treatment will be given for 50 minutes in each session. Electrical muscle stimulation (EMS) will be applied in prone lying before every session of hypopressive exercises (HE). A device will use for muscle stimulation at 7Hz for 15 minutes. The intensity of current will gradually increase from zero to a minimum that can be tolerated by the patient. Two electrodes will place medially to the ischial tuberosity and the remaining two will place on the sacral area.
  After a 2-minute interval, the patient will be asked to perform HE in an upright position. For this maneuver, the patient will be instructed to inhale, then breathe to expand the ribcage, and then exhale completely. Hold the breath out before relaxing core and ribcage. Four sets of 10 repetitions with a 3-minute interval between each set will be performed.
  Interventions: Other: Hypopressive exercises
- Pelvic floor muscle exercises and electrical muscle stimulation (EMS) (Experimental): Women included in this group underwent 24 sessions during 8 weeks (3 days/ week). Treatment will be given for 50 minutes in each session. Electrical muscle stimulation (EMS) will be applied in prone lying before every session of pelvic floor muscle exercises. A device will use for muscle stimulation at 7Hz for 15 minutes. The intensity of current will gradually increase from zero to a minimum that can be tolerated by the patient. Two electrodes will place medially to the ischial tuberosity and the remaining two will place on the sacral area.
  After a 2-minute interval, the patient will be asked to perform pelvic floor muscle exercises in a sitting position. The patient is instructed to hold each contraction for 6 seconds, with three to four contractions added on the top. Four sets of 10 repetitions with a 2-minute interval between each set will be performed.
  Interventions: Other: Pelvic floor exercises

INTERVENTIONS:
Other: Hypopressive exercises — For hypopressive exercises, the patient will be instructed to inhale, then breathe to expand the ribcage, and then exhale completely. Hold the breath out before relaxing core and ribcage.
  Arms: Hypopressive exercises and electrical muscle stimulation (EMS)
Other: Pelvic floor exercises — For pelvic floor exercises, the patient is instructed to hold each contraction for 6 seconds.
  Arms: Pelvic floor muscle exercises and electrical muscle stimulation (EMS)

SUMMARY:
The aim of our study is to compare the effects of hypopressive exercises with routine pelvic floor exercises in improving the frequency and severity of urinary incontinence in women and also to enhance their quality of life as it worsens after childbirth, pregnancy, and in older age.

DETAILED DESCRIPTION:
A randomized control trial study will be conducted in which patients with urinary incontinence will be assigned to group 1 that will receive hypopressive exercises with electrical muscle stimulation (EMS) and patients in group 2 will receive pelvic floor exercises with EMS.

The intervention will be applied (3 days/week) for 8 weeks. Four sets of 10 repetitions with a 3-minute interval between each set will be performed for group 1 in an upright position while four sets of 10 repetitions with a 2-minute interval between each set will be performed for group 2 in the sitting position.

ELIGIBILITY:
Inclusion Criteria:

* Women aged between 20 to 65 years
* Gynecologist and urologist diagnosed patients
* Participants not engaged systematically in sports or physical activities(≤ sessions per week, ≤ weeks per week)

Exclusion Criteria:

* If participants had hypertension or any serious mental disease
* Pregnancy or up to 2 months postpartum
* Urge fecal incontinence or vaginal pain
* Underwent any physiotherapy for urinary incontinence before
* Any kidney disease

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2022-02-20 (Actual); Study Completion 2022-02-20 (Actual)

PRIMARY OUTCOMES:
International Consultation Incontinence Questionnaire Short Form (ICIQ-SF) | 8th week
  ICIQ-SF is a screening tool for incontinence. 4 main items (a total of 6) ask for a rating of symptoms in past four weeks. Item 1 and 2 are demographics so items 3,4,5 are summed for a total score. Using a score value, UI is classified as mild (1-5), moderate (6-12), severe (13-18), very severe (19-21) from a total score ranges from 0-21.
International Impact Questionnaire, Short Form (IIQ-7) | 8th week
  IIQ-7 is a reliable tool for measuring the impact on quality of life for UI patients. Calculate the mean of all items and then subtract the mean by 1, then multiply by 100/3 (0-100 range).
Medical, Epidemiologic and Social aspects of Aging Questionnaire (MESA Questionnaire) | 8th week
  It is a reliable and validated tool to evaluate the severity and predominance of stress and urge urinary incontinence. The MESA Questionnaire consists of 15 items total divided into stress (1-9) and urge (10-15) subscales. The total score of urgency (18) and stress (27) is divided into three degrees. For urgency, a score of 1-6 is categorized as mild, 7-12 moderate, and 13-18 as severe. For stress, a score of 1-9 is categorized as mild, 10-18 moderate, and 19-27 as severe. A higher MESA score indicates more frequent symptoms overall ranges from 0-45.

CONTACTS AND LOCATIONS:
Overall Officials: Muhmmad Kashif, Study Chair — Riphah International University
Locations (1):
- Riphah International University, Faisalābad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No